CLINICAL TRIAL: NCT05101473
Title: Exercise Therapy for People With a Diabetic Foot Ulcer - a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exercise for DFU; REG-075-2021 (Other: Datatilsynet); SJ-928 (Other: Videnskabsetisk Komite)
Record Dates: First submitted 2021-10-18; First posted 2021-11-01 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Wound Healing Disorder; Ulcer Foot; Ulcer Healing
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The trial is a single-center single-group feasibility trial in outpatient clinical settings.
  The trial will be reported with reference to the extended CONSORT guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise therapy (Experimental): Exercises will be performed with minimal weight bearing on foot soles, as recommended in the literature for people with diabetic peripheral neuropathy.
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Exercise Therapy — The overall framework will consist of two supervised exercise sessions per week of 30-60 min duration for 12 weeks in order to be able to result in the physiological adaptions that are needed to improve the health of the individual participant.

SUMMARY:
The aim of this feasibility study is to evaluate a 12-week exercise intervention in people with an active diabetic foot ulcer through pre-defined research progression criteria (participant recruitment and retention, duration of the collection of outcome measures, adherence to the exercise programme, and adverse events), besides participant and physiotherapist feedback, self-reported outcomes and objective measurements in preparation for a potential future RCT.

The primary study hypothesis is that exercise therapy for people with an active diabetic foot ulcer will have high participant recruitment and adherence to treatment and that it does not affect wound healing negatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* Diabetes mellitus
* Non-surgical ulcer located distal to the malleoli
* Willingness to participate in a 12-week supervised exercise therapy intervention twice a week
* Prescribed with a therapeutic shoe, orthopaedic specialist shoe from the outpatient clinic or a specialized podiatrist.

Exclusion Criteria:

* Dementia or other reasons that cause inability to give informed consent
* People that are wheelchair-bound
* People with a prescribed cast or walker boot
* Unable to understand Danish.
* Diagnosed with or awaiting evaluation of suspected acute phase Charcot arthropathy or osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 month
  will be analysed by dividing number of included participants (n = 15) by the number of months it took to include them (calculated from study start until the 15th participant is recruited).
Participant retention | 12-week follow up.
  will be evaluated by the number of participants showing up at 12-week follow up.
Exercise adherence | 12-week follow up.
  will be evaluated using exercise logs completed at each session by the physiotherapist covering load and intensity. Adherence will be calculated by counting number of exercise sessions completed in the exercise log, divided by 24 planned sessions, presented in percentage.
Adverse events | 12-week follow up.
  Safety will be assessed based on observed and patient-reported adverse events, and their relatedness to the index ulcer and to the exercise program.
  Minor adverse events will cover muscle soreness or post-exercise fatigue. Whereas serious adverse events will cover all negative events related to the foot ulcer, and cover life- threatening events, disability, or permanent damage
Participant and physiotherapist feedback | 12-week follow up.
  will be provided at 12-week follow up on a custom-made interviews with open questions on acceptability of assessment procedures, treatment experience, and feedback about the supervised sessions and potential adverse events
30-second chair-stand test | 12-week follow up.
  To test leg strength and endurance of participants the 30-second chair-stand test will be performed at baseline and at the last day of follow-up.
Tandem Test | 12-week follow up.
  Balance will be evaluated with the Tandem Test at baseline and at the last day of follow-up.
Ulcer size | 12-week follow up.
  Ulcer size measurement is assessed on digital images with standardized measuring tape from participants last to the outpatient clinic visit prior to baseline and from participants last to the outpatient clinic visit to last day of follow-up. The measurement is a standard measurement in the outpatient clinic at every participant visit
Wound-QoL | 12-week follow up.
  Participants are asked to fill out the the Wound-QoL questionnaires in paper form at baseline and at the last day of follow-up
  The Wound-QoL consists of 17 items that can be combined into three individual multi-item domains: Body, Psyche and Everyday life as well as a single-item domain on Economy
EC-5D-5L | 12-week follow up.
  Participants are asked to fill out the Danish versions of the patient-reported outcome measures (PROM) EQ-5D-5L in paper form at baseline and at the last day of follow-up.
  The EQ-5D- 3L includes the European Quality of life visual analogue scale (EQ-VAS) where the patient's own health 'today' is rated between 0 (worst imaginable health) and 100 (best imaginable health)
4x10-meter fast-paced walk test | 12-week follow up.
  The 40 m FPWT is a test for performance on the activity short-distance walking. The test will be performed at baseline and at the last day of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- SUH Køge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Undecided